CLINICAL TRIAL: NCT00735176
Title: Treatment of Cervical Radiculopathy With Arthroplasty Compared With Discectomy With Fusion and Cage (ACDF. Clinical, Radiological and Biomechanical Aspects. A Randomized Multicenter Study.
Brief Title: The Norwegian Cervical Arthroplasty Trial
Acronym: NORCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Rikshospitalet University Hospital (Other); Haukeland University Hospital (Other); Ullevaal University Hospital (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.2008.211 (REK); 18809/2/AMS (Other: NSD)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Radiculopathy, Cervical
Keywords: Radiculopathy, cervical; Nerve Root Compression; Disc, intervertebral; Intervertebral Disk Displacement; Spondylosis; Spinal Osteophytosis; Arthroplasty, replacement; Diskectomy; Spinal Fusion
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement; Spondylosis; Spinal Osteophytosis | interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artificial Cervical Disc (Experimental): Anterior cervical discectomy, followed by insertion of the Discover™ Artificial Cervical Disc
  Interventions: Procedure: Cervical arthroplasty
- ACDF (Active Comparator): Anterior cervical discectomy and fusion (ACDF)
  Interventions: Procedure: Anterior cervical discectomy and fusion (ACDF)

INTERVENTIONS:
Procedure: Cervical arthroplasty — Anterior cervical discectomy, followed by insertion of the Discover™ Artificial Cervical Disc
  Other Names: Discover™ Artificial Cervical Disc
  Arms: Artificial Cervical Disc
Procedure: Anterior cervical discectomy and fusion (ACDF) — Anterior cervical discectomy and decompression, followed by insertion of a PEEK cage, which induces fusion.
  Other Names: Cage is made of polyetheretherketone (PEEK)
  Arms: ACDF

SUMMARY:
The study will compare cervical arthroplasty with cervical discectomy and fusion, in the treatment of cervical radiculopathy. The 0-hypothesis is that there is no difference between the two methods, when comparing primary and secondary outcome variables.

DETAILED DESCRIPTION:
Anterior discectomy and fusion (ACDF) is in Norway currently the most common operative method against cervical radiculopathy, caused by disc herniation and/or spondylosis. In the last decade cervical arthroplasty has emerged as a new alternative operative method. Arthroplasty is claimed to preserve the natural motion of the spine, thereby preventing adjacent level disc disease and providing better clinical results. However, this hypothesis has not yet been adequately proven. In our study, we will prove if there is any real difference in terms of clinical effect between cervical arthroplasty and ACDF.We will also compare the overall costs of the two methods, including cost-utility analyses. Moreover, we will study the development of adjacent level disease by use of MRI scans, and analyze cervical spine motion and disc height by use of Distortion Compensated Roentgen Analysis (DCRA).

ELIGIBILITY:
Inclusion Criteria:

* Age 25 - 60 years
* Clinical C6 or C7 root radiculopathy with corresponding radiologic findings with or without neurological symptoms
* Mechanical provoked pain which aggravate with physical activity or positive Spurling test
* Radiological nerve root compression on the basis of disc herniation or spondylosis
* NDI =/> 30 percent
* The patient has not responded to non-operative treatment and shown no sign of improvement during the last 6 weeks

Exclusion Criteria:

* Significant spondylosis involving more than one level
* Intramedullary changes on MRI
* Ankylosis at adjacent level
* Clinical suspicion of myelopathy
* Chronic generalised pain syndrome
* Infection
* Active cancer
* Rheumatoid arthritis involving the cervical spine
* Previous trauma involving the cervical spine
* Pregnancy
* Allergy against contents in cage/artificial disc
* Previous neck surgery
* Psychological or somatic illness that causes the patient not to be suitable for the study
* The patient does not understand Norwegian orally or in writing.
* Abuse of medication/narcotics

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
change in Neck Disability Index (NDI) | up to 5 years

SECONDARY OUTCOMES:
Clinical effect, measured by use of EQ5-D, SF-36, numeric arm/neck pain registration, dysphagia score, rate of complications/reoperations/morbidity | Preoperatively. Postoperatively: 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years
Health economical aspects, measuring hospital costs, patient costs, primary health service costs, and performing cost-utility analyses. | Postoperatively: 3 months, 6 months, 1 year, 2 years
Adjacent level disc disease, measured by use of MRI scans. | Maximum 4 months preoperatively. Postoperatively:1 year, 2 years, 5 years
Preservation of cervical translational and rotational segmental motion, disc height and dorsoventral displacement, by use of functional X-rays with Distortion Compensated Roentgen Analysis (DCRA) | Preoperatively. Postoperatively: 1 day, 6 weeks, 1 year, 2 years, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Øystein P Nygaard, Professor MD, Study Chair — Department of Neurosurgery, St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Sundseth J, Jacobsen EA, Kolstad F, Sletteberg RO, Nygaard OP, Johnsen LG, Pripp AH, Andresen H, Fredriksli OA, Myrseth E, Zwart JA. Heterotopic ossification and clinical outcome in nonconstrained cervical arthroplasty 2 years after surgery: the Norwegian Cervical Arthroplasty Trial (NORCAT). Eur Spine J. 2016 Jul;25(7):2271-8. doi: 10.1007/s00586-016-4549-6. Epub 2016 Apr 9. PMID 27061727
- [Result] Sundseth J, Fredriksli OA, Kolstad F, Johnsen LG, Pripp AH, Andresen H, Myrseth E, Muller K, Nygaard OP, Zwart JA; NORCAT study group. The Norwegian Cervical Arthroplasty Trial (NORCAT): 2-year clinical outcome after single-level cervical arthroplasty versus fusion-a prospective, single-blinded, randomized, controlled multicenter study. Eur Spine J. 2017 Apr;26(4):1225-1235. doi: 10.1007/s00586-016-4922-5. Epub 2016 Dec 23. PMID 28012081
- [Derived] Johansen TO, Sundseth J, Fredriksli OA, Andresen H, Zwart JA, Kolstad F, Pripp AH, Gulati S, Nygaard OP. Effect of Arthroplasty vs Fusion for Patients With Cervical Radiculopathy: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2119606. doi: 10.1001/jamanetworkopen.2021.19606. PMID 34351401